CLINICAL TRIAL: NCT06172777
Title: A Study to Evaluate the Consistency of Oscillometry and Spirometry Test Results in Patients With Confirmed or Suspected Asthma or COPD
Acronym: IOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589BR00078
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Asthma/ COPD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- suspected asthma: enrollment 200 subjects
  Interventions: Diagnostic Test: suspected asthma
- Suspected COPD: enrollment 200 subjects
  Interventions: Diagnostic Test: suspected COPD
- confirmed asthma: enrollment 200 subjects
  Interventions: Diagnostic Test: confirmed asthma
- confirmed COPD: enrollment 200 subjects.
  Interventions: Diagnostic Test: confirmed COPD

INTERVENTIONS:
Diagnostic Test: suspected asthma — enrollment 200 asthma patients
  Groups: suspected asthma
Diagnostic Test: suspected COPD — enrollment 200 COPD patients
  Groups: Suspected COPD
Diagnostic Test: confirmed asthma — enrollment 200 patients
  Groups: confirmed asthma
Diagnostic Test: confirmed COPD — enrollment 200 patients
  Groups: confirmed COPD

SUMMARY:
The study to evaluate the consistency of oscillometry and spirometry test results in patients with confirmed or suspected asthma or COPD, it is a multi-centre clinical study. sponsor by Astrazeneca Investment(China) Co.,LTD.

DETAILED DESCRIPTION:
800 patients, including suspected or confirmed asthma, suspected or confirmed COPD, will be enrolled in nationwide multiple study centres. Enrolling suspected and confirmed subject in an approximate1:1 rate in centre-level. About 100 subjects were enrolled at the leader site, while about 14 subjects were enrolled at other sites.

To evaluate the consistency of oscillometry and spirometry test results in patients with confirmed or suspected asthma or COPD.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply and signed informed content :

Suspected and confirmed asthma

1. Participant must be≥18 years old.
2. Present symptom such as wheezing, cough, chest tightness, shortness of breath, but not confirmed-asthma (without evidence of variable airflow restriction) or confirmed-asthma with evidence of variable airflow restriction (such as positive bronchodilation test, positive bronchial challenge test, variability >10% in twice daily PEF over 2 weeks, et al) Suspected and confirmed COPD

1 Participant must be ≥40 years old. 2 Present symptom such as chronic cough, sputum production, dyspnoea, but not confirmed-COPD (without evidence of persistent airflow restriction) or confirmed- COPD with evidence of persistent airflow restriction (post-bronchodilator FEV1/FVC<0.7)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Any diseases that influence lung function result such as lung cancer, pneumonia, active pulmonary tuberculosis, pulmonary embolism and interstitial lung disease, etc; history of recent surgery that affect lung function results, including thoracotomy surgery, pneumothorax surgery, thoracic drainage, etc
2. Contraindication to spirometry or oscillometry test, or allergic to bronchodilator.
3. Currently pregnant or breast-feeding women
4. Judge by the investigator if the participant is unlikely to comply with study procedures, restrictions, and requirements, will not be enrolled .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected and confirmed adult asthma and COPD patients.
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Kappa coefficient of normal result and abnormal result between oscillometry and spirometry pre-BDT in the overall population. | 30Dec2024
  The consistency between oscillometry and spirometry results pre-bronchodilator test (BDT) in overall population.

SECONDARY OUTCOMES:
Compare the time required from attempting to complete the test and number of attemptsB before completing the test. | 30Dec2024
  To compare the physician and patient acceptability to complete the first test of oscillometry and spirometry
Kappa coefficient of bronchodilator test positive result C between oscillometry and spirometry in the overall population. | 30Dec2024
  To evaluate the bronchodilator test result consistent of oscillometry with spirometry in overall population
Kappa coefficient of normal result and abnormal result between oscillometry and spirometry post-BDT in COPD group. | 30Dec2024
  The consistency between oscillometry and spirometry post-BDT results in COPD group

OTHER OUTCOMES:
Characteristics of the population with consistent / inconsistent results from oscillometry and spirometry in BDT. | 30Dec2024
  To explore the characteristics of populations with consistent results between oscillometry and spirometry
To explore the correlation of Asthma Control Questionnaire (ACQ-5) scores with spirometry and oscillometry parameters. | 30Dec2024
  To explore the parameters which can reflect asthma control better between oscillometry and spirometry in asthma patients
To explore the correlation of modified Medical Research Council (mMRC) scores with spirometry and oscillometry parameters | 30Dec2024
  To explore the parameters which can correlates better with symptom between oscillometry and spirometry in COPD patients
The predict value of oscillometry parameters including R5, R5-R20,X5, AX, fres, DX5 (X5 intra-breath) and DAX (AX intra-breath) pre bronchodilator test in differentiate between asthma and COPD | 30Dec2024
  To explore the predict value of oscillometry parameters includingR5, R5-R20, X5, AX, fres, DX5 (X5 intra-breath) and DAX (AX intra-breath) pre-bronchodilator test in differentiation between asthma and COPD
The consistency between oscillometry parameters (R5, R5-R20,X5, AX fres) (normal,mild, moderate, severe)and FEV1 %pred(≤30%;30%-50%;50%-80%;≥80%) in preBDT | 30Dec2024
  To explore consistency between oscillometry parameters (R5, R5-R20,X5, AX fres) (normal,mild, moderate, severe)and FEV1 %pred(≤30%;30%-50%;50%-80%;≥80%) in pre-BDT
The consistency between oscillometry parameters (R5, R5-R20,X5, AX fres) (normal,mild, moderate, severe)and FEV1 %pred(≤30%;30%-50%;50%-80%;≥80%) in post BDT. | 30Dec2024
  To explore consistency between oscillometry parameters (R5, R5-R20,X5, AX fres) (normal,mild, moderate, severe)and FEV1 %pred(≤30%;30%-50%;50%-80%;≥80%) in post BDT
To identify the joint predictors with the best diagnostic values for the diagnosis of COPD/asthma | 30Dec2024
  To identify the best joint predictors for the diagnosis of COPD/asthma
To explore the characteristics of patients with small airway dysfunction defined by oscillometry and spirometry, and whether they are agreeing in detecting small airway dysfunction. | 30Dec2024
  To describe the characteristics of patients with small airway dysfunction using spirometry and oscillometry in the overall population, as well as the Kappa coefficient for detect small airway dysfunction between oscillometry and spirometry.
To explore the SAE/medical device deficiency related to ALDS or the investigational procedure | 30Dec2024
  SAE/medical device deficiency related to ALDS or the investigational procedure

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Fengcheng
  - Research Site, Fuyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hanchuan
  - Research Site, Hangzhou
  - Research Site, Haozhou
  - Research Site, Henan
  - Research Site, Hong Kong
  - Research Site, Jinan
  - Research Site, Jingzhou
  - Research Site, Kunming
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Ordos
  - Research Site, Panzhou
  - Research Site, Qionghai
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Suining
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Xinyang
  - Research Site, Yulin
  - Research Site, Yunnan
  - Research Site, Zhaotong
  - Research Site, Zhengzhou
  - Research Site, Zhuji
  - Research Site, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BR00078&attachmentIdentifier=4380bb7a-694e-4278-8b10-bd35fa3ab570&fileName=D589BR00078_IOS_synopsis__V1.0_20250331.pdf&versionIdentifier=